CLINICAL TRIAL: NCT03266978
Title: Impact of the Glycemic State on the in Hospital and Short Term Outcomes of Patients With ST-segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Angioplasty
Brief Title: Impact of Glycemic State on Patients ST Elevation Myocardial Infarction With Primary Percutaneous Coronary Angioplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, El shaimaa Abd El Fattah Omran, pricipal investgator, Assiut University
Other Study IDs: ODMI Assiut
Record Dates: First submitted 2017-08-24; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ST-elevation myocardial infarction is a major cause of morbidity and mortality worldwide. ST-elevation myocardial infarction damages the regional myocardium that undergoes ischemia and necrosis, resulting in impairment of both systolic and diastolic functions of the heart. Left ventricular function and myocardial infarct size both serve as the main determinants Of patients' outcome after myocardial infarction. Timely management of ST-elevation myocardial infarction, using reperfusion therapy, including fibrinolysis and primary percutaneous coronary intervention, leads to a better outcome for these patients.

DETAILED DESCRIPTION:
Reperfusion failure is attributed to different factors, including diabetes. Several mechanisms have been proposed for the harmful effects of hyperglycemia after acute myocardial infarction. Association of hyperglycemia with the activation of blood coagulation has been well studied; it could induce a shortening of the fibrinogen half-life, increase in fibrinopeptide A, fragments of pro-thrombin in factor VII, and platelet aggregation, all of which could lead to increased activation of thrombosis. Hyperglycemia at admission is associated with increased levels of inflammatory markers, enhanced expression of cytotoxic T-cells, and reduced expression of cytotoxic T-lymphocyte-associated protein 4, indicating its association with increased inflammatory immune process after acute myocardial infarction. It also could be associated with endothelial dysfunction, oxidative stress, and possibly, abolition of protective ischemic preconditioning. Other possible mechanism of harmful effects of acute hyperglycemia is microvascular dysfunction after coronary revascularization.

Studying the influence of diabetes mellitus on clinical outcome in the thrombolytic era of acute myocardial infarction, GUSTO-I trial showed that patients with diabetes mellitus have a significantly increased risk of both early and late mortality, which may be attributed to more advanced coronary artery disease and co-morbidities.

Results of the HORIZONS-AMI study showed that patients with newly diagnosed diabetes mellitus had similarly poor prognosis after primary percutaneous coronary intervention in ST-elevation myocardial infarction patients as those with previously established diabetes mellitus, newly diagnosed diabetes mellitus was based on HgbA1c levels following admission and did not assess for blood glucose levels at admission or during hospital stay.

Regarding the effect of diabetes mellitus on left ventricular systolic function, diabetic patients with first ST-elevation myocardial infarction had reduced left ventricular systolic function, measured with speckle-tracking strain, compared with non-diabetic patients at baseline and at 6-month follow up, despite similar left ventricular ejection fraction in both groups. Similarly, according to the ischemic cascade, diastolic function is expected to be affected with variable degrees among diabetic, prediabetic and non-diabetic ST-elevation myocardial infarction patients.

Timmer et al, studied the effect of admission stress hyperglycemia and that of chronic hyperglycemia (elevated levels of HbA1c in patients with undiagnosed diabetes mellitus) on ST-elevation myocardial infarction patients undergoing primary percutaneous coronary intervention; both elevated glucose and HbA1c levels were associated with adverse outcomes. However elevated glucose but not elevated HbA1c was associated with larger enzymatic infarct size and high early mortality.

Furthermore, Ota et al, demonstrated the association between stress hyperglycemia and the development of microvascular obstruction using late gadolinium enhancement - cardiovascular magnetic resonance imaging, suggesting that hyperglycemic control immediately after admission might reduce the incidence of microvascular obstruction.

This study is designed to explore the impact of the glycemic state on the in-hospital and short term outcomes of patients with ST-elevation myocardial infarction undergoing reperfusion therapy in two separate arms; those with known diabetes mellitus and those without known diagnosis of diabetes mellitus, and then comparing results among those with controlled diabetes mellitus, uncontrolled diabetes mellitus and newly diagnosed diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* The study will be performed on acute ST-elevation myocardial infarction patients with/without history of diabetes mellitus undergoing primary percutaneous coronary intervention.

Exclusion Criteria:

* Patients not treated with primary percutaneous coronary intervention.
* Patients with prior myocardial infarction, prior primary percutaneous coronary intervention and/or coronary artery bypass graft (altering disease state).
* Patients with cardiogenic shock (altering disease state).
* Patients with severe liver or renal disease (altering disease state).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting to investigators Coronary Care Unit - Assiut University Heart Center with acute ST-elevation myocardial infarction undergoing primary percutaneous coronary intervention.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Admission glucose level | Baseline .
  Blood glucose level on admission measured by mmol/l .

SECONDARY OUTCOMES:
To evaluate left ventricular systolic function. | Baseline and latter at 6 months follow-up.
  Using transthoracic echocardiography.
To evaluate left ventricular diastolic function. | Baseline and latter at 6 months follow-up.
  Using transthoracic echocardiography.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ertelt K, Brener SJ, Mehran R, Ben-Yehuda O, McAndrew T, Stone GW. Comparison of Outcomes and Prognosis of Patients With Versus Without Newly Diagnosed Diabetes Mellitus After Primary Percutaneous Coronary Intervention for ST-Elevation Myocardial Infarction (the HORIZONS-AMI Study). Am J Cardiol. 2017 Jun 15;119(12):1917-1923. doi: 10.1016/j.amjcard.2017.03.016. Epub 2017 Mar 29. PMID 28427734
- [Result] Ota S, Tanimoto T, Orii M, Hirata K, Shiono Y, Shimamura K, Matsuo Y, Yamano T, Ino Y, Kitabata H, Yamaguchi T, Kubo T, Tanaka A, Imanishi T, Akasaka T. Association between hyperglycemia at admission and microvascular obstruction in patients with ST-segment elevation myocardial infarction. J Cardiol. 2015 Apr;65(4):272-7. doi: 10.1016/j.jjcc.2014.10.013. Epub 2014 Dec 19. PMID 25533423
- [Result] Iwakura K. Stress hyperglycemia and microvascular obstruction after acute myocardial infarction. J Cardiol. 2015 Apr;65(4):270-1. doi: 10.1016/j.jjcc.2014.11.012. Epub 2014 Dec 29. No abstract available. PMID 25553870
- [Result] Marfella R, Siniscalchi M, Esposito K, Sellitto A, De Fanis U, Romano C, Portoghese M, Siciliano S, Nappo F, Sasso FC, Mininni N, Cacciapuoti F, Lucivero G, Giunta R, Verza M, Giugliano D. Effects of stress hyperglycemia on acute myocardial infarction: role of inflammatory immune process in functional cardiac outcome. Diabetes Care. 2003 Nov;26(11):3129-35. doi: 10.2337/diacare.26.11.3129. PMID 14578250
- [Result] Sattur S, Sarwar B, Sacchi TJ, Brener SJ. Correlation between markers of reperfusion and mortality in ST-elevation myocardial infarction: a systematic review. J Invasive Cardiol. 2014 Nov;26(11):587-95. PMID 25364000